CLINICAL TRIAL: NCT02512913
Title: Family Smoking Cessation in Romania Using Pregnancy as a Window of Opportunity
Acronym: QuitTogether
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Cristian Meghea, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: K01TW009654 (NIH)
Record Dates: First submitted 2015-07-10; First posted 2015-07-31 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Tobacco Smoking; Pregnancy
Keywords: Smoking Cessation; Intervention; Pregnancy; Postnatal
MeSH Terms: conditions — Tobacco Smoking; Smoking Cessation | interventions — Acclimatization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted/enhanced MAPS (Experimental): Counseling sessions delivered by phone to the pregnant/postpartum women and to the husbands/partners
  Interventions: Behavioral: Adapted/enhanced MAPS
- Usual Care (No Intervention): Couples in the control condition will receive usual care

INTERVENTIONS:
Behavioral: Adapted/enhanced MAPS — The plan is for recruitment at the first prenatal care visit followed by a proposed eight-session phone counseling sequence for the women, consistent with the session frequency in the original MAPS intervention: 1st call at 14 weeks gestation (75% of Romanian women begin prenatal care in 1st trimester), three monthly calls through the 2nd trimester (18-22-26 weeks gestation), a 5th and 6th calls in the 3rd trimester (32 and 36 weeks), and two postnatal calls (2 and 6 weeks postpartum). Four calls are planned for the partners: at 14-, 22-, and 32-weeks, and at 2-weeks postpartum.
  Arms: Adapted/enhanced MAPS

SUMMARY:
The purpose of this research is to adapt and implement a pregnancy and postnatal smoking cessation intervention for couple that will begin early in pregnancy and have an additional postnatal component.

DETAILED DESCRIPTION:
Pregnancy smoking and postnatal relapse are highly prevalent in Romania and Central and Eastern Europe, with lifetime negative health effects for the women and their children. There are higher odds of female smoking persistence during pregnancy, and of relapse once pregnant women quit, when the male partner also smokes.

Building on ongoing pilot work led by Dr. Meghea with Babes-Bolyai University (BBU) in Cluj-Napoca, Romania, the overall objective of the proposed research, conducted through BBU in the same target population as the ongoing pilot, is to adapt, enhance, and test the implementation feasibility and preliminary efficacy of an evidence-based pregnancy and postnatal couple intervention for smoking cessation that begins early in pregnancy and has a postnatal component.

The intervention will be based on the motivation and problem solving (MAPS) approach, successful in preventing smoking relapse postpartum in the US, which will be enhanced by targeting the couples' smoking behavior by focusing on dyadic efficacy for smoking cessation. The target population is primigravida pregnant women and their partners in Cluj-Napoca, Romania.

The specific aims are: (1) To develop an adapted and enhanced couple intervention to reduce pregnancy smoking and postpartum relapse in Romania based on the MAPS approach. (2) To conduct a pilot randomized controlled trial to test the fidelity of the culturally adapted MAPS intervention enhanced for couples smoking prevention during pregnancy and postpartum. (3) To examine in the pilot the implementation feasibility and initial efficacy in increasing maternal pregnancy smoking cessation and reducing postnatal relapse, with secondary hypotheses regarding maternal smoking reduction and spousal cessation, relapse, and reduction.

This study will form the basis for a larger, multicenter clinical trial that will be submitted by Dr. Meghea as an R01 application by the end of the 4th year of this award to evaluate the effectiveness of the proposed smoking prevention intervention. If proven effective in the subsequent R01 trial, the intervention has a high potential for broad spectrum population impact and sustainability. The long-term goal is the adoption in the national Romanian health system as a proactive extension of the existing STOP SMOKING national program which includes a quitline.

ELIGIBILITY:
Inclusion Criteria:

* the woman is pregnant,
* she is a smoker
* 18 years or older (legal age for consent and for consuming tobacco in Romania)
* married or in a stable relationship
* phone service in the home or mobile phone
* willing to have the partner contacted for participation, upon brief explanation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
maternal smoking abstinence (questionnaire, biochemical verified) | assessments at recruitment, at 32-weeks during pregnancy, and at 16 weeks after birth
  assessed at multiple time points during the project

SECONDARY OUTCOMES:
maternal smoking abstinence (questionnaire) | assessments at recruitment, at 32-weeks during pregnancy, and 16 weeks after birth
  assessed at multiple time points during the project

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Meghea, PhD, Principal Investigator — Michigan State University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania